CLINICAL TRIAL: NCT06152315
Title: Study of Splay Sign in Mitral Regurgitation and Other Valve Lesions as Related to Its Mechanisms, Predictors of Its Occurence and Association With Severity of Mitral Regurgitation
Brief Title: Mitral Splay Sign, Its Mechanism and Association With Severity of Regurgitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ITMO University (Other)
Responsible Party: Principal Investigator, Artemiy Okhotin, researcher in Digital Public Health Technologies, ITMO University
Other Study IDs: TARUSA SPLAY STUDY
Record Dates: First submitted 2023-10-30; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Mitral Regurgitation
Keywords: echocardiography; splay sign; seagull cry
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mitral splay sign: Patients with at least mild mitral regurgitation and splay sign on color doppler echocardiography
- no mitral splay sign: Patients with at least mild mitral regurgitation and no splay sign on color doppler echocardiography

SUMMARY:
To study echocardiography splay sign in mitral regurgitation and its association with mitral regurgitation severity and doppler band artifact ('seagull cry').

ELIGIBILITY:
Inclusion Criteria:

* any patient undergoing echocardiography for clinical indications

Exclusion Criteria:

* poor quality of recorded echocardiography study
* inability to ascertain severity of mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to echocardiography in community hospital in Tarusa
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Presence of mitral splay sign | 1 year
  Logical, Presence of splay sign -- wide linear color doppler artifact on the level of valve coaptation disproportional to the width of the regurgitant jet
Presence of narrow doppler bands | 1 year
  Logical, presence of narrow bands during continuous doppler echocardiography assessed by two echocardiographers (one blinded)

SECONDARY OUTCOMES:
Mitral regurgitation severity | 1 year
  Categorical, Grade of severity of mitral regurgitation assessed by echocardiography by two independent echocardiographers

OTHER OUTCOMES:
Blood pressure | 1 year
  Numerical, Arterial blood pressure measured during the study
Age | 1 year
  Numerical, Age of the patient
Gender | 1 year
  Categorical, Gender of the patient
BMI | 1 year
  Numerical, Body mass index (weight divided by squared height)

CONTACTS AND LOCATIONS:
Locations (1):
- Tarusa Hospital, Tarusa, Kaluga Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
All the data including anonymized echocardiography studies.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: along with the publication
Access Criteria: publicly accessible